CLINICAL TRIAL: NCT04726436
Title: The Impact of Timing and Dosing of Dextrose Solution on Postoperative Nausea and Vomiting.
Brief Title: Dextrose Effect on Postoperative Nausea and Vomiting (PONV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dextrose PONV
Record Dates: First submitted 2021-01-24; First posted 2021-01-27 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Glucose; Water; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dextrose 5% (Experimental): 100 mL/ hour of dextrose 5% were given starting 1 hour before operation and continue till approximately middle of surgery by communicating with surgeon to assess the timing and dosing of dextrose solution effect on PONV.
  Interventions: Other: Dextrose 5% in water
- Dextrose 10% (Experimental): 100 mL/ hour of dextrose 10% were given starting 1 hour before operation and continue till approximately middle of surgery by communicating with surgeon
  Interventions: Other: Dextrose 10%
- Saline placebo (Placebo Comparator): 100 mL/ hour of normal saline were given starting 1 hour before operation and continue till approximately middle of surgery by communicating with surgeon
  Interventions: Other: Saline placebo

INTERVENTIONS:
Other: Dextrose 5% in water — One hour before operation, patients were given dexrose 5%100/hour only for 2 hours to end at about middle of surgery
  Arms: Dextrose 5%
Other: Dextrose 10% — One hour before operation, patients were given dexrose 10 %100/hour only for 2 hours to end at about middle of surgery
  Arms: Dextrose 10%
Other: Saline placebo — One hour before operation, patients were given normal saline100/hour only for 2 hours to end at about middle of surgery
  Other Names: Normal saline
  Arms: Saline placebo

SUMMARY:
The aim of this study to assess which time and dose of dextrose solution more effective in decreasing postoperative nausea and vomiting.

DETAILED DESCRIPTION:
All patients signed informed consent after excluding patients not candidate for the study.patients were divided to three groups, taking either 0.9% saline as control group(group C), dextrose 5%(group D5) or dextrose 10%(group D10).

ELIGIBILITY:
Inclusion Criteria:

* Female non-smokers adults (age 18-65 years)
* ASA I-II who were listed for elective surgery under general anesthesia (surgery which is risk for PONV).

Exclusion Criteria:

* Severe hypertension
* Coagulopathy
* Significant hepatic or renal disease
* Diabetes mellitus or abnormal blood glucose on the morning of surgery
* Withdrawal of consent
* Severe intraoperative hypotension requiring large volume intravascular fluid treatment
* Protocol violations including nitrous oxide administration.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting within 24 hour | 24hour after surgery
  Number of participants who experienced PONV grade ≥2 as assessed by PONV score . The PACU nurses assessed and documented PONV using a Verbal Descriptive Scale, which correlates to visual analog nausea scores, with an objective measure of severity: 0 = no PONV: patient reports no nausea and has had no emesis episodes; 1 = mild PONV: patient reports nausea but declines antiemetic treatment; 2 = moderate PONV: patient reports nausea and accepts antiemetic treatment; and 3 = severe PONV: nausea with any emesis episode (retching or vomiting). The score was obtained at 0, 30, 60, 90, and 120 minutes after PACU arrival; thus 5 scores were recorded during PACU stay. A 24-hour PONV assessment that elicited any nausea and emesis episode since PACU discharge was obtained by a blinded investigator by telephone or in person at the patient's bedside (delayed PONV).

SECONDARY OUTCOMES:
Number of doses of antiemetics required to control PONV. | 24hour postoperative
  Frequency of doses of antiemetics required to control postoperative nausea and vomiting, initial antiemetic treatment was 10 mg slow IV metoclopramide for occurred nausea or 4 mg IV ondansetron for occurred nausea & vomiting or if the previous treatment failed for nausea
Number of classes of antiemetics | 24 hour postoperative
  Frequency of classes of antiemetics required to control postoperative nausea and vomiting, Initial antiemetic treatment was 10 mg slow IV metoclopramide for occurred nausea or 4 mg IV ondansetron for occurred nausea & vomiting or if the previous treatment failed for nausea

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zorrilla-Vaca A, Marmolejo-Posso D, Stone A, Li J, Grant MC. Perioperative Dextrose Infusion and Postoperative Nausea and Vomiting: A Meta-analysis of Randomized Trials. Anesth Analg. 2019 Oct;129(4):943-950. doi: 10.1213/ANE.0000000000004019. PMID 30649067